CLINICAL TRIAL: NCT05255796
Title: Influence of Different Intraocular Lenses on IOL-capsular Complex After Cataract Surgery in Patients With High Myopia: a Clinical Observation Based on SS-OCT
Brief Title: IOL-capsular Complex After Different Intraocular Lenses Implantation in Patients With High Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20211213CTR
Record Dates: First submitted 2021-12-13; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Age-related Cataract
Keywords: High Myopia; Various Types of IOLs; The position of IOL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-piece (Experimental): The patients' axial length is over 26 mm and are diagnosed age related cataract or complicated cataract.
  Interventions: Procedure: one-piece
- plate-haptic (Experimental): The patients' axial length is over 26 mm and are diagnosed age related cataract or complicated cataract.
  Interventions: Procedure: plate-haptic

INTERVENTIONS:
Procedure: one-piece — Patients underwent phacoemulsification cataract surgery with one-piece IOL implantation.
  Arms: one-piece
Procedure: plate-haptic — Patients underwent phacoemulsification cataract surgery with plate-haptic IOL implantation.
  Arms: plate-haptic

SUMMARY:
The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation. Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity. IOL decentration ≥ 0.4 mm or/and IOL tilt ≥7degree were considered clinically significant cause of poor post-surgery visual quality especially for optical sophisticated IOLs. This negative impact does not affect various types of IOLs equally. Several studies indicated that AL was an independent risk factor of IOL decentration and tilt for emmetropic or moderate myopic eyes. For patients with high myopia, they often have a longer axial length and a larger capsule diameter, which reduces the rotational stability of the IOL and may lead to tilt, decentration and displacement of IOL. Currently, there is no literature guidance to compare the results of cataract surgery combined various types of IOLs implantation in patients with high myopia. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can evaluate the IOL capsule bending and the lens position after cataract surgery. Also, CASIA2 can be used to documented the dynamic changes of IOL-capsular complex after surgery.

DETAILED DESCRIPTION:
The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation. Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity. Although up to 2-3 degree tilt and a 0.2-0.3 mm decentration are common and clinically unnoticed for any design of IOL, larger extent of tilt and decentration has a negative impact on the optical performance. IOL decentration ≥ 0.4 mm or/and IOL tilt ≥7degree were considered clinically significant cause of poor post-surgery visual quality especially for optical sophisticated IOLs. This negative impact does not affect various types of IOLs equally. Several studies indicated that AL was an independent risk factor of IOL decentration and tilt for emmetropic or moderate myopic eyes. However, there is scarce evidence on characteristics and factors associated with clinically significant IOL decentration and tilt in highly myopic eyes. For patients with high myopia, they often have a longer axial length and a larger capsule diameter, which reduces the rotational stability of the IOL and may lead to tilt, decentration and displacement of IOL. Currently, there is no literature guidance to compare the results of cataract surgery combined various types of IOLs implantation in patients with high myopia. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can evaluate the IOL capsule bending and the lens position after cataract surgery. Also, CASIA2 can be used to documented the dynamic changes of IOL-capsular complex after surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed age related cataract or complicated cataract with axial length over 26mm
* The patients' age over 18 years old
* The patients plan to receive cataract surgery in Eye hospital of Wenzhou Medical University
* The dialated pupils are over 6mm
* Patients are willing and able to complete the follow-ups

Exclusion Criteria:

* Patients with other types of cataract
* Patients have complications in the surgery and after surgery
* Patients have other severe diseases of eyes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The position of IOL | The 1st day after surgery
  Evaluation of the position of IOL through tilt, decentration and the process of capsule bending using CASIA2.
The position of IOL | The 1st week after surgery
  Evaluation of the position of IOL through tilt, decentration and the process of capsule bending using CASIA2.
The position of IOL | The 1st month after surgery
  Evaluation of the position of IOL through tilt, decentration and the process of capsule bending using CASIA2.
The position of IOL | The 3rd month after surgery
  Evaluation of the position of IOL through tilt, decentration and the process of capsule bending using CASIA2.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Eye Hospital of Wenzhou Medical College, Hangzhou, Zhejiang, China